CLINICAL TRIAL: NCT03944642
Title: Breastfeeding as a Health-promoting Behavior: Design and Piloting of a Complex Intervention to Support Breastfeeding Self-efficacy: CRIAA Program
Brief Title: Design and Piloting of a Complex Intervention to Support Breastfeeding Self-efficacy (CRIAA Program)
Acronym: CRIAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: University of Navarra (Other)
Responsible Party: Principal Investigator, Camila Lucchini, Associate Professor, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PIEM04-19
Record Dates: First submitted 2019-05-03; First posted 2019-05-09 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Breastfeeding; Self Efficacy
Keywords: Complex Intervention; Pilot Study; Breastfeeding Support
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Masking Description: The allocation was done by outpatient clinic to avoid contamination bias. Participants of the outpatient clinic A will receive the CRIAA Program (intervention group) and participants of the outpatient clinic B will receive the standard care (control group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive the standard prenatal care and invited to participate of a breastfeeding workshop during the third trimester of pregnancy, with active and intentional participation of the pregnant woman and her partner/relative; based on adult education methodology. In addition, women participants will have continuous support during their breastfeeding process, up to 6 months of the child's life, through a virtual support group (whats-app), where they will receive messages that promote their self-efficacy in relation to their ability to breastfeed and may ask questions that are related to breastfeeding. Professionals in this group will be train before delivering the intervention.
  Interventions: Behavioral: Breastfeeding support
- Standard Care (No Intervention): This group will receive the standard pre and postnatal regular care, for mother and child. Professionals who provide direct care will maintain their usual attention.

INTERVENTIONS:
Behavioral: Breastfeeding support — Breastfeeding self-efficacy enhancing through professional support
  Other Names: CRIAA Program
  Arms: Intervention

SUMMARY:
The aim of the study is to design and pilot the effect of a complex intervention to support mothers' breastfeeding self-efficacy and professional self-efficacy to support breastfeeding families, considering breastfeeding as a health promoting behavior. Specific objectives are the evaluation of feasibility and acceptability of the intervention, and estimate the preliminary effect on maternal and professional self-efficacy.

DETAILED DESCRIPTION:
Breastfeeding is the optimal feeding during early childhood. However, the prevalence of exclusive breastfeeding is not as expected. The evidence of effectiveness of interventions designed to support breastfeeding is not conclusive. Breastfeeding is a complex experience, influenced by numerous factors, as self-efficacy, that require interdisciplinary approaches.The aim of the study is to design and pilot the effect of a complex intervention to support mothers' breastfeeding self-efficacy and professional self-efficacy to support breastfeeding families, considering breastfeeding as a health promoting behavior. The project will be done in two stages a) design of the intervention and b) experimental pilot trial with control and intervention groups, for evaluation of feasibility, acceptability of the intervention and preliminary estimate of its effect on maternal and professional self-efficacy. The project will be carry out in two public outpatient clinics (Centro de Salud Familiar Alberto Hurtado y Centro de Salud Familiar Juan Pablo II) in Santiago, Chile. Participants will be breastfeeding women and their partner/family member; and health professionals who provide care to mother and child. Intervention group will receive a breastfeeding workshop during the third trimester of pregnancy and on-line breastfeeding support during the first 6 months postpartum. Health professionals will be train to deliver the intervention.Control group will receive the standard care as provided in the outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* Being in physiological pregnancy in the third trimester
* Speak Spanish
* Give informed consent

Exclusion Criteria:

* Pathology during pregnancy that entails difficulties for breastfeeding
* Multiple pregnancy
* Breastfeeding especial situations (cleft lip and palate, congenital heart disease and newborn's hospitalization)
* Preterm birth (at <37 weeks gestation)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Mothers self-efficacy: spanish validated version of Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) | At five points: week 28 - 40 pregnancy (T1); and 10 days (T2); 2 months (T3); 4 months (T4); and 6 months (T5) after birth
  Changes on maternal breastfeeding self-efficacy using the Spanish validated version of Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF). BSES-SF is a 14 item, unidimensional, self-report instrument developed to measure a mother's confidence in her ability to breastfeed. All items are presented with a 5-point Likert-type scale where 1 indicates "not at all confident" and 5 indicates "always confident" (scores: minimum 14 and maximum 70). Higher scores indicate higher levels of breastfeeding self-efficacy.
Professionals self-efficacy in relation to their ability to support breastfeeding mothers: APCLA Scale (Professional Self Efficacy for Breastfeeding Care Scale) | At three points: before professional training (the same day that the intervention begins) (T1); 3 months (T2) and 6 months (T3) after the beginning of the intervention
  Changes on professional self-efficacy in relation to their ability to support breastfeeding mothers using the Professional Self Efficacy for Breastfeeding Care Scale (Autoeficacia Profesional para los Cuidados en Lactancia, APCLA). APCLA scale is a 14 item, unidimensional, self-report instrument developed to measure a professional's confidence in her/his ability to support a breastfeeding mother. All items are presented with a 5-point Likert-type scale where 1 indicates "not at all confident" and 5 indicates "always confident" (scores: minimum 14 and maximum 70). Higher scores indicate higher levels of breastfeeding support self-efficacy. This scale was constructed and validated in Spanish based on the Spanish version of BSES-SF

SECONDARY OUTCOMES:
Proportion of participants mothers/mothers invited to participate (Feasibility) | Baseline
  Proportion of participants mothers/mothers invited to participate to measure the recruitment process of the CRIAA program
Duration in minutes of the breastfeeding workshop (Feasibility) | Baseline
  Duration in minutes of the breastfeeding workshop (scheduled time v/s time used) to measure the implementation of the CRIAA program
Participants recruitment. Participants that complete the intervention/total of participants recruited (Feasibility) | At two times: Baseline (T1) and at the end of the intervention at 6 moths of age of the child (T2)
  Participants that complete the CRIAA Program/total of participants recruited to measure participant's retention of the CRIAA program
Acceptability of the intervention by mothers | At six months of age of the child, when intervention is over
  Explored by semi-structured interviews, without using any scale. The script of the interviews will contain questions about positive and negative aspects of the program perceived by participant mothers
Acceptability of the intervention by professionals | At two times: Three months post intervention begins by semi-structured interviews (T1) and when study is over, an average of 10 months, by a focus group (T2)
  Explored by semi-structured interviews and focus group with professionals
Acceptability of participation in decision making by mothers and their partner/relative | At five points: week 28 - 40 pregnancy (T1); and 10 days (T2); 2 months (T3); 4 months (T4); and 6 months (T5) after birth
  Changes on perceived participation in decision making related to the child's type of feeding, using the Spanish validated version of CollaboRate. It is a short and self-applying generic instrument that allows measuring user participation in a particular health decision (Cronbach's alpha> 0.89). It consists of three questions with alternative answers with a likert scale of 1 to 7. In this project, both the mothers and the partner /relative will be asked about their participation in the decision to feed the child. The version that will be used is validated in Chilean population (CollaboRate Chile)

OTHER OUTCOMES:
Breastfeeding percentage | At four times: 10 days (T1), 2 months (T2), 4 months (T3), and 6 months (T4)
  Percentage of children with exclusive breastfeeding

CONTACTS AND LOCATIONS:
Overall Officials: Camila Lucchini-Raies, MSc,BSc,RN, Principal Investigator — Profesor Asociado Escuela de Enfermeria Pontificia Universidad Catolica de Chile
Locations (4):
- Chile (3):
  - Escuela de Enfermeria Pontificia Universidad Catolica de Chile, Santiago
  - Centro de Salud Familiar ANCORA San Alberto Hurtado, Santiago
  - Centro de Salud Familiar ANCORA Juan Pablo II, Santiago
- Facultad de Enfermeria Universidad de Navarra, Pamplona, Spain

REFERENCES:
- [Derived] Lucchini-Raies C, Marquez-Doren F, Perez JC, Campos S, Beca P, Lopez-Dicastillo O. A complex intervention to support breastfeeding: A feasibility and acceptability study. Int J Nurs Pract. 2023 Dec;29(6):e13184. doi: 10.1111/ijn.13184. Epub 2023 Jul 18. PMID 37461904
- [Derived] Lucchini-Raies C, Marquez-Doren F, Beca P, Perez JC, Campos S, Lopez-Dicastillo O. The CRIAA Program complex intervention in primary care to support women and their families in breastfeeding: Study protocol for a pilot trial. J Adv Nurs. 2020 Dec;76(12):3641-3653. doi: 10.1111/jan.14534. Epub 2020 Oct 15. PMID 33058232